CLINICAL TRIAL: NCT04406558
Title: Psychological Impact of the Health Measures Generated by the SarsCov-2 Pandemic in Adolescents (COVADO)
Brief Title: Psychological Impact of the Health Measures Generated by the COVID19 in Adolescents
Acronym: COVADO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: COVADO
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Psychological Adaptation; Psychology, Social
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — An online questionnaire on the experience of the period of confinement and deconfinement will be sent to the cohort of adolescents followed at the CHI Creteil for a chronic disease or not. Forty adolescents will be randomly selected for a remote interview on the experience and memorization of the period of confinement and deconfinement.
  Other Names: Interview

SUMMARY:
The lockdown of the French population is a health measure put in place in response to the pandemic linked to a new coronavirus, SARS-CoV-2 (Covid-19). After a health campaign to recommend hygienic "barrier gestures" and social distancing, the decision to confine the population at the national level was decided by the executive from Monday 16 March to Monday 11 May 2020. The national confinement implies the restriction of movement to the strict necessary, outings near the home and the closure of schools and communities. These decisions have led to an unprecedented state of stress for the entire French population, the consequences of which are unknown in the short, medium or long term. The objectives of this study are to evaluate the psychological impact of the confinement on adolescents with or without chronic disease and also the difficulties and fears engendered by deconfinement .

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 11 to 18 years old
* Previous consultation in the Centre Hospitalier intercommunal de Creteil
* Agree to participate

Exclusion Criteria:

* Lack of computer equipment or internet connection

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be proposed to all the adolescents followed in the Centre hospitalier Intercommunal de Creteil for a chronic disease or not.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Anxiety score from the Generalized Anxiety Disorder 7 (GAD-7) questionnaire | At inclusion
  Scale 0-21

SECONDARY OUTCOMES:
Depression score from the Adolescent Depression Rating Scale (ADRS) questionnaire | At inclusion
  Scale 0-60
Post traumatic score questionnaire: Children's Revised Impact of Events Scales -CRIES13 | At inclusion
  8 items that are scored on a four-point scale and 3 sub scales: intrusion (4 items); avoidance (4 items) and arousal (5 items)
Presence or absence of difficulty in falling asleep, sleeping | At inclusion
  a question on the quality and quantity of sleep will be asked to the teenager on a questionnaire
Presence or absence of feeding difficulty | At inclusion
  a question on the presence or absence of feeding difficulty will be asked to the teenager on a questionnaire
Presence or absence of difficulty performing physical activity | At inclusion
  a question on the presence or absence of difficulty performing physical activity will be asked to the teenager on a questionnaire
Presence or absence of toxic consomption (drug, acohol) during the lockdown | At inclusion
  a question on the presence or absence of toxic consomption will be asked to the teenager on a questionnaire
Mean duration time in front of screen (hours per day) | At inclusion
Presence or absence of difficulties with social interactions | At inclusion
  A question on the presence or absence of difficulties with social interactions will be asked to the teenager on a questionnaire
Presence or absence of difficulties with familial interactions | At inclusion
  Presence or absence of difficulties with familial interactions

CONTACTS AND LOCATIONS:
Locations (1):
- Camille JUNG, Créteil, France